CLINICAL TRIAL: NCT04659226
Title: MicroRNA Profile in Women With Migraine Before and After Treatment With Erenumab
Brief Title: MicroRNA Profile and Erenumab Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Simona Sacco, Full Professor of Neurology, University of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAMG334AIT05T
Record Dates: First submitted 2020-11-05; First posted 2020-12-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Migraine
Keywords: cgrp; monoclonal antibodies; microRNA; epigenetic; migraine prevention
MeSH Terms: conditions — Migraine Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Episodic or chronic migraine (Experimental): Women starting treatment with erenumab according to clinical indication
  Interventions: Genetic: Blood sampling for microRNA testing

INTERVENTIONS:
Genetic: Blood sampling for microRNA testing — Blood samples will be collected and analyzed for the microRNA profile by means of microfluidic cards

SUMMARY:
Erenumab, a monoclonal antibody acting on the calcitonin gene-related peptide (CGRP) receptor, is an effective and safe migraine-specific preventive drug. The use of migraine-specific preventive drugs paves the way for a novel method to study migraine pathogenesis. Migraine is a complex disorder with several genetic and epigenetic influence, including that of microRNA. Several microRNAs, including those of inflammation and of endothelial function, have high expression levels in subjects with migraine; however, the findings of the available studies are insufficient to provide epigenetic biomarkers for migraine. Besides, little evidence is available on the role of migraine preventive treatments in the expression of microRNA. The study aims at evaluating the expression profiles of microRNAs before and after erenumab treatment prescribed according to clinical indication. The study will include women with episodic or chronic migraine treated with erenumab 140 mg monthly according to the Summary of Product Characteristics and local reimbursement criteria. The study will compare the expression profile of microRNAs in women with episodic and chronic migraine; besides, it will investigate differences in migraine-associated microRNA expression according to age, migraine characteristics, pain intensity, response to erenumab, migraine-related impact and disability.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 50 years
* Chronic or episodic migraine with or without aura diagnosed according to the International Classification of Headache Disorders - 3rd edition
* Receiving a first prescription of erenumab for migraine prevention according to the Summary of Product Characteristics and local reimbursement criteria
* At least 1 year from migraine onset
* Provided informed consent

Exclusion Criteria:

* Headache other than migraine
* Prior exposure to erenumab or other monoclonal antibodies targeting CGRP or its receptor
* Use of any migraine preventive treatment in the last 60 days or 5 half-lives or 4 months if ever treated with botulinum toxin A
* Pregnant or nursing
* Body Mass Index <18 or >30 Kg/m2
* Heavy smoking (more than 20 cigarettes per day)
* Myocardial infarction, stroke, transient ischemic attack, unstable angina, or coronary artery bypass surgery or other revascularization procedures within 12 months prior to first visit
* Illicit drug abuse
* Major psychiatric disorders
* Infective or inflammatory diseases
* Any chronic medication prescribed for indications different from migraine within 60 days before study initiation

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Fold changes in microRNA serum concentration - Episodic migraine | 3 months per each patient
  Relative quantification of circulating microRNAs expression changes in women with episodic migraine after a 3-month treatment with erenumab with respect to pre-treatment. Data will be obtained by real-time polymerase chain reaction on microfluidic cards. Details on tested microRNAs are provided at the following link: https://assets.thermofisher.com/TFS-Assets/GSD/Reference-Materials/tac-advanced-miRNA-assay-list.xlsx
Fold changes in microRNA serum concentration - Chronic migraine | 3 months per each patient
  Relative quantification of circulating microRNAs expression changes in women with chronic migraine after a 3-month treatment with erenumab with respect to pre-treatment. Data will be obtained by real-time polymerase chain reaction on microfluidic cards. Details on tested microRNAs are provided at the following link: https://assets.thermofisher.com/TFS-Assets/GSD/Reference-Materials/tac-advanced-miRNA-assay-list.xlsx

SECONDARY OUTCOMES:
Baseline comparison between episodic and chronic migraine | Baseline
  Relative quantification of microRNA expression levels at baseline in women with chronic compared with episodic migraine. Data will be obtained by real-time polymerase chain reaction on microfluidic cards. Details on tested microRNAs are provided at the following link: https://assets.thermofisher.com/TFS-Assets/GSD/Reference-Materials/tac-advanced-miRNA-assay-list.xlsx
Subgroup analyses | 3 months per each patient
  Subgroup analyses of patients stratified according to age, migraine characteristics, response to erenumab, and migraine-related impact and disability. Data will be obtained by real-time polymerase chain reaction on microfluidic cards. Details on tested microRNAs are provided at the following link: https://assets.thermofisher.com/TFS-Assets/GSD/Reference-Materials/tac-advanced-miRNA-assay-list.xlsx

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ornello R, Zelli V, Compagnoni C, Caponnetto V, De Matteis E, Tiseo C, Tessitore A, Sacco S. MicroRNA profiling in women with migraine: effects of CGRP-targeting treatment. J Headache Pain. 2024 May 16;25(1):80. doi: 10.1186/s10194-024-01787-2. PMID 38755568